CLINICAL TRIAL: NCT03987854
Title: The University of Michigan PCOS Intervention Using Nutritional Ketosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Laura Saslow, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00113697; P30DK092926 (NIH); K01DK107456 (NIH)
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Results first posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Polycystic Ovary Syndrome
Keywords: nutrition
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Participants will be taught how to follow a very low carbohydrate, ketogenic diet, become more physically active, and get adequate sleep. Behavioral: positive affect informational materials. They will also be taught about positive affect skills, such as gratitude, positive reappraisal, and personal strengths, in addition to information about mindfulness and mindful eating techniques.
Masking Description: Laboratory results will be assessed by a lab not associated with the study team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- complete diet and lifestyle program (Experimental)
  Interventions: Behavioral: diet and lifestyle program

INTERVENTIONS:
Behavioral: diet and lifestyle program — Participants will be taught how to follow a very low carbohydrate, ketogenic diet, become more physically active, and get adequate sleep. They will also be taught taught about positive affect skills (such as gratitude, positive reappraisal, and personal strengths) and mindfulness (general mindfulness and mindful eating).

SUMMARY:
The goal of this proposal is to pilot test our existing very-low carbohydrate diet intervention, adapted for women with PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a common and costly ($4.3 billion/year) endocrine disorder that significantly impairs quality of life and increases the risk of obesity and type 2 diabetes as well as hyperandrogenism, infertility, hyperlipidemia, and cardiovascular disease. Diet and lifestyle weight-loss interventions are recommended as the first-line treatment of PCOS, but experts disagree about which nutritional approach is best. A review of previous diet and lifestyle trials in PCOS did find a slight benefit of lower carbohydrate diets for weight loss, glucose control, insulin, and insulin resistance. This may be because carbohydrate intake leads to increased insulin secretion, which then stimulates ovarian androgen production and inhibits the release of fatty acids from cells, both of which worsen PCOS-related issues. Although lower carbohydrate diets may be helpful, research from other populations with or at risk of type 2 diabetes suggests that prior PCOS studies may have set insufficient carbohydrate reduction targets. The investigators propose that a very-low carbohydrate diet may be needed to especially benefit women with PCOS, as greater carbohydrate reduction should have a larger impact on androgen levels and weight loss. Thus, the goal of this proposal is to pilot test our existing very-low carbohydrate diet intervention, adapted for women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* We will include women in one PCOS subtype, those having these two symptoms:

  * Hyperandrogenism - (a) If not on current birth control: hyperandrogenism defined as current elevated total testosterone >= 50 ng/dL or free androgen index > 1.5 (ratio of testosterone/SHBG x 100) or severe acne or hirsutism (b) if on current birth control: history from the past 10 years of hyperandrogenism defined as past elevated total testosterone >= 50 ng/dL or free androgen index > 1.5 (ratio of testosterone/SHBG x 100) or severe acne or hirsutism
  * oligomenorrhea-anovulation defined as spontaneous intermenstrual periods of ≥ 45 days or a total of ≤ 8 menses per year.

Participants must also be:

* overweight or obese (BMI 25-50)
* be 21-40 years old
* have regular access to the internet
* be able to engage in light physical activity
* willing and able to follow the assigned intervention.

Exclusion Criteria:

* a non-English speaker
* inability to complete baseline measurements
* a substance abuse, mental health, or medical condition that would interfere with participation (such as current chemotherapy)
* pregnant or planning to get pregnant in the next 6 months
* type 1 or type 2 diabetes
* baseline aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2 times normal
* baseline renal disease defined as BUN > 30 mg/dL or serum creatinine >1.4 mg/dL
* baseline uncorrected thyroid disease (TSH <0.45 mIU/ML or >4.5 mIU/ML)
* breastfeeding or less than 6 months post-partum
* planned or history of weight loss surgery
* vegan or vegetarian
* currently enrolled in a weight loss program or other investigative study that might conflict with this research
* taking medications known to cause weight gain or loss
* taking hypoglycemic medications other than metformin or medications known to affect metabolism
* or patients with other etiologies of anovulation and hyperandrogenism, e.g., Cushing's disease, thyroid dysfunction, elevated prolactin levels, signs of congenital adrenal hyperplasia, organic intra cranial lesion such as a pituitary tumor, or suspected adrenal or ovarian tumor secreting androgens.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on sex.
Enrollment: 29 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Missel AL, O'Brien AV, Maser H, Kanwal A, Bayandorian H, Martin S, Carrigan P, McNamee R, Daubenmier J, Isaman DJM, Padmanabhan V, Smith YR, Aikens JE, Saslow LR. Impact of an online multicomponent very-low-carbohydrate program in women with polycystic ovary syndrome: a pilot study. F S Rep. 2021 Sep 4;2(4):386-395. doi: 10.1016/j.xfre.2021.08.008. eCollection 2021 Dec. PMID 34934978

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Complete Diet and Lifestyle Program
Started | 29
Completed | 21
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: all participants at baseline
Arm/Group | Complete Diet and Lifestyle Program
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.21 (5.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 24
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Body Weight Loss
Description: Mean percent body weight loss was defined as: (weight at 4 months - baseline weight) / (baseline weight) *100.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: percentage of weight
Arm/Group | Complete Diet and Lifestyle Program
Number analyzed (Participants) | 21
percentage of weight | -7.67 (6.10)
Statistical Analysis 1: Comparison: Complete Diet and Lifestyle Program; Test type: Superiority; p < .001, t-test, 2 sided — -6.16; paired t-test = -7.67, Standard Deviation 6.10

2. Secondary Outcome: HbA1c Change
Description: percentage of glycosylated hemoglobin
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: units of %
Arm/Group | Complete Diet and Lifestyle Program
Number analyzed (Participants) | 21
units of % | -0.21 (0.27)
Statistical Analysis 1: Comparison: Complete Diet and Lifestyle Program; Test type: Superiority; p = .001, t-test, 2 sided — -3.29; paired t-test = -0.21, Standard Deviation 0.27

3. Other Pre Specified Outcome: Polycystic Ovary Syndrome Questionnaire (PCOSQ): Emotions
Description: Scale measures health-related quality-of-life for Women with PCOS with five domains: emotions, body hair, weight, infertility, and menstrual problems. It is a 7-point scale questionnaire assessing health-related quality of life specific to PCOS in 5 different domains, with "7" representing optimal function and "1" representing poorest function.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Complete Diet and Lifestyle Program
Number analyzed (Participants) | 21
score on a scale | 1.92 (1.17)
Statistical Analysis 1: Comparison: Complete Diet and Lifestyle Program; Test type: Superiority; p < .001, t-test, 2 sided — 7.52; paired t-test = 1.92, Standard Deviation 1.17

4. Other Pre Specified Outcome: Polycystic Ovary Syndrome Questionnaire (PCOSQ): Body Hair
Description: as for outcome 3
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Complete Diet and Lifestyle Program
Number analyzed (Participants) | 21
score on a scale | 1.14 (1.04)
Statistical Analysis 1: Comparison: Complete Diet and Lifestyle Program; Test type: Superiority; p < .001, t-test, 2 sided — 5.03; paired t-test = 1.14, Standard Deviation 1.04

5. Other Pre Specified Outcome: Polycystic Ovary Syndrome Questionnaire (PCOSQ): Weight
Description: as for outcome 3
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Complete Diet and Lifestyle Program
Number analyzed (Participants) | 21
score on a scale | 2.52 (1.70)
Statistical Analysis 1: Comparison: Complete Diet and Lifestyle Program; Test type: Superiority; p < .001, t-test, 2 sided — 6.81; paired t-test = 2.52, Standard Deviation 1.70

6. Other Pre Specified Outcome: Polycystic Ovary Syndrome Questionnaire (PCOSQ): Infertility
Description: as for outcome 3
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Complete Diet and Lifestyle Program
Number analyzed (Participants) | 21
score on a scale | 1.08 (1.43)
Statistical Analysis 1: Comparison: Complete Diet and Lifestyle Program; Test type: Superiority; p = .003, t-test, 2 sided — 3.46; paired t-test = 1.08, Standard Deviation 1.43

7. Other Pre Specified Outcome: Polycystic Ovary Syndrome Questionnaire (PCOSQ): Menstrual Symptoms
Description: as for outcome 3
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Complete Diet and Lifestyle Program
Number analyzed (Participants) | 21
score on a scale | 1.11 (1.56)
Statistical Analysis 1: Comparison: Complete Diet and Lifestyle Program; Test type: Superiority; p = .004, t-test, 2 sided — 3.26; paired t-test = 1.11, Standard Deviation 1.56

8. Other Pre Specified Outcome: Polycystic Ovary Syndrome Questionnaire (PCOSQ): Menstrual Predictability
Description: as for outcome 3
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Complete Diet and Lifestyle Program
Number analyzed (Participants) | 21
score on a scale | 2.10 (2.76)
Statistical Analysis 1: Comparison: Complete Diet and Lifestyle Program; Test type: Superiority; p = .002, t-test, 2 sided — 3.49; paired t-test = 2.10, Standard Deviation 2.76

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Complete Diet and Lifestyle Program
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 3/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Complete Diet and Lifestyle Program (N=29)
kidney stones (Renal and urinary disorders) | 2 — Two participants developed kidney stones, one within 2 weeks of starting the intervention and the other 2 months into the intervention.
blurry vision (Eye disorders) | 1 — A participant reported continuous muscle cramping and blurry vision 2 months into the intervention; symptoms subsided after consulting with their physician.
muscle cramping (Musculoskeletal and connective tissue disorders) | 1 — A participant reported continuous muscle cramping and blurry vision 2 months into the intervention; symptoms subsided after consulting with their physician.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/54/NCT03987854/Prot_SAP_001.pdf
  • Informed Consent Form (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT03987854/ICF_002.pdf